CLINICAL TRIAL: NCT00824954
Title: Evaluation of Extracorporeal Photochemotherapy in Children and Young Adults With Refractory Acute Graft Versus Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Extracorporeal Photopheresis in Children and Young Adults With Refractory Acute Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Etienne MERLIN, CHU Clermont-Ferrand
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0043
Record Dates: First submitted 2008-12-18; First posted 2009-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Graft Versus Host Disease
Keywords: 0 to 30 years; Refractory Acute GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Eosinophil Cationic Protein

INTERVENTIONS:
Procedure: ECP (performed on Themos UVAR-XTS or external UVA irradiator after cell collection by apheresis) — ECP (performed on Thermos UVAR-XTS or external UVA irradiator after cell collection by apheresis)

SUMMARY:
Purpose : to evaluate the efficacy of ECP in children with refractory acute GVHD This study addresses patients with persistent GVHD after steroid and/or monoclonal antibody therapy

DETAILED DESCRIPTION:
One arm. Six sessions in two weeks. Classification in complete response (resolution of all signs of GVHD), partial response (improvement of at least one grade) or absence of response (Glucksberg criteria). Tapering depending on patient condition during weeks 2 to 10. Final evaluation at week 10. Steroid therapy tapering at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 30 years
* Acute GVHD refractory to steroids (disease progression after 2 days or absence of response after 4 days) and/or second line therapy (absence of response after 8 days)
* patient consent and/or parent consent

Exclusion Criteria:

* less of 10 kgs BW
* clinical or biological state precluding the apheresis
* previous GVHD therapy with anti-lymphocyte serum (excepted in the conditioning regimen)

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
GVHD grading | during weeks 2 to 10

SECONDARY OUTCOMES:
Overall survival Incidence of chronic GVHD | during weeks 2 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Merlin, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France